CLINICAL TRIAL: NCT01501279
Title: Ultrasound Guided Pudendal Block in Transurethral Prostatectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, consultant MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Diskapi2011
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2011-12

CONDITIONS: Pain, Postoperative
Keywords: pudendal nerve block; postoperative pain; bladder spasm
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pudendal nerve block (Experimental): USG guided pudendal nerve block performed under general anesthesia
  Interventions: Procedure: Pudendal nerve block
- no nerve block (No Intervention): Control group without nerve block

INTERVENTIONS:
Procedure: Pudendal nerve block — the pudendal nerve block is going to be performed to the medial of ischial tuberosity with USG guidance in lithotomy position
  Arms: pudendal nerve block

SUMMARY:
The pudendal nerve conveys sensory, motor, sympathetic fibres to the perineum, bladder neck and proximal urethra. Pain management during transurethral procedures is a major concern.Patients who have been catheterized under anesthesia complained of urgency in the postoperative period because of catheter-related bladder irritation. We want to investigate that the effect of pudendal block to postoperative pain, bladder spasm and patient comfort in transurethral prostatectomies

DETAILED DESCRIPTION:
Outcome measures USG guided transperineal pudendal block success Postoperative pain score (VAS score) Postoperative bladder spasm (Severity of bladder discomfort will record as severe(behavioral responses such as strong vocal response, flailing limbs),moderate (not accompanied by any behavioral responses) and no bladder discomfort.

Postoperative patient's comfort (poor, sufficient, good)

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II,III status
* Who were scheduled to have elective transurethral resection of the prostate

Exclusion Criteria:

* Chronic renal failure
* coagulopathy
* active anorectal disease
* active urinary tract infection
* uncontrolled diabetes

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
postoperative bladder spasm | postoperative 12 h
  Postoperative bladder spasm (Severity of bladder discomfort will record as severe(behavioral responses such as strong vocal response, flailing limbs),moderate (not accompanied by any behavioral responses) and no bladder discomfort.

SECONDARY OUTCOMES:
postoperative pain | postoperative 12 h
  VAS score (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Derya Özkan, MD, Principal Investigator — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic; Taylan Akkaya, MD, Study Director — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic; Nihat Karakoyunlu, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Urology Clinic; Julide Ergil, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. AnesthesiologyClinic; Hamit Ersoy, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 3. Urology Clinic
Locations (1):
- Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic, Ankara, Turkey (Türkiye)